CLINICAL TRIAL: NCT01867515
Title: Spectral Dynamics and Speech Understanding by Hearing Impaired People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C1020-R; 5I01RX001020-03 (NIH)
Record Dates: First submitted 2013-05-20; First posted 2013-06-04 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Hearing; Hearing Loss, sensorineural; Speech Perception
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Younger normally-hearing listeners (Active Comparator): Participants with auditory thresholds within the normal limits.
  * age between 18 and 35
  * individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz Acoustic distortion of speech
  Interventions: Other: Acoustic distortion of speech
- Hearing-impaired listeners (Active Comparator): individuals with bilateral sensorineural hearing losses with thresholds between 25 and 70 dB HL and no losses greater than 70 dB HL at frequencies of 4000 Hz or below
  * age 18 to 65 Acoustic distortion of speech
  Interventions: Other: Acoustic distortion of speech
- Older normally-hearing listeners (Active Comparator): Participants with auditory thresholds within the normal limits.
  * age between 36 and 65
  * individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz Acoustic distortion of speech
  Interventions: Other: Acoustic distortion of speech

INTERVENTIONS:
Other: Acoustic distortion of speech

SUMMARY:
The purpose of this program of research is to understand the perception of the dynamic spectral properties of speech by hearing-impaired listeners, with the long-term goal of improving speech understanding by these individuals in adverse listening conditions. The proposed research compares the performance of normally-hearing and hearing-impaired listeners on measures of speech understanding in the presence of different types of signal distortion and speech understanding of signals with enhanced spectral dynamics. A computational model based on the amount of potential information available in speech will be used to quantify differences in speech intelligibility due to hearing status and stimulus characteristics.

DETAILED DESCRIPTION:
This is a behavioral study of human auditory perception. Each experiment in this study involves prospective data collection from three types of listeners. The experimental listeners will be people with sensorineural hearing loss and the control listeners will either be subjects with normal hearing or normal-hearing listeners for whom hearing loss will be simulated through the use of a spectrally-shaped broadband noise. The tasks of the subjects in this study involve either listening to synthesized sounds over earphones while seated comfortably in a sound-treated booth, and making responses indicating the subject's auditory perception of these sounds by touching specific areas on a touch-screen terminal; or, listening to recorded, acoustically modified syllables, words, or sentences over earphones and making responses indicating the subject's identification.

ELIGIBILITY:
Inclusion Criteria:

* individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz
* or, individuals with bilateral sensorineural hearing losses with thresholds between 25 and 70 dB HL and no losses greater than 70 dB HL at frequencies of 4000 Hz or below

Exclusion Criteria:

* a conductive hearing impairment or other otological pathology
* hearing thresholds greater than 70 dB HL at any frequencies of 4000 Hz or below or pure-tone averages (averaged across 500, 1000, and 2000 Hz) of greater than 65 dB HL
* bilateral differences greater than 20 dB at any frequency below 4000 Hz
* an inability to complete the experimental tasks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Molis, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Younger Normally-hearing Listeners: Participants with auditory thresholds within the normal limits.
  * age 18 to 35
  * individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz
- Older Normally-hearing Listeners: Participants with auditory thresholds within the normal limits.
  * age 36 to 65
  * individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz
- Hearing-impaired Listeners: individuals with bilateral sensorineural hearing losses with thresholds between 25 and 70 dB HL and no losses greater than 70 dB HL at frequencies of 4000 Hz or below
  * age 18 to 65
Period: Overall Study
Arm/Group | Younger Normally-hearing Listeners | Older Normally-hearing Listeners | Hearing-impaired Listeners
Started | 13 | 12 | 25
Completed | 13 | 11 | 14
Not Completed | 0 | 1 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Younger Normally-hearing Listeners | Older Normally-hearing Listeners | Hearing-impaired Listeners | Total
Number analyzed (Participants) | 13 | 11 | 14 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 13 | 36
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 26.5 [20 to 33] | 59.1 [51 to 65] | 59.4 [48 to 65] | 48.0 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 2 | 13
  Male | 7 | 6 | 12 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percent Correct Words Identified
Description: The experimental approach compares speech identification performance among younger, normally-hearing listeners, older normally-hearing listeners and hearing-impaired listeners. Tasks will be carried out in quiet and in the presence of continuous, speech-shaped background noise. The investigators compared the understanding of unprocessed stimuli with 1) time-compressed stimuli, 2) time-compressed stimuli expanded in time via gaps and 3) uncompressed stimuli where portions of the signal were replaced with silence. Experimental metrics were percentage of correct/incorrect speech identification in each listening condition.
Time Frame: average of two blocks per condition obtained over the course of up to three 2-hour visits, spaced an average of one week apart
Measure: Mean (Full Range); unit: percentage of words identified
Groups:
- Normally-hearing Listeners: Participants with auditory thresholds within the normal limits.
  * age 18 to 35
  * individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz
- Older Normally-hearing: Participants with auditory thresholds within the normal limits.
  * age 36 to 65
  * individuals with hearing thresholds of 20 dB HL or better at all octave frequencies between 250 Hz and 4000 Hz
- Hearing-impaired Listeners: individuals with bilateral sensorineural hearing losses with thresholds between 25 and 70 dB HL and no losses greater than 70 dB HL at frequencies of 4000 Hz or below
Arm/Group | Normally-hearing Listeners | Older Normally-hearing | Hearing-impaired Listeners
Number analyzed (Participants) | 13 | 11 | 14
percentage of words identified
  Unprocessed speech in quiet | 98.6 [88 to 100] | 97.1 [84 to 100] | 91.9 [64 to 100]
  Unprocessed speech in noise | 98.8 [88 to 100] | 96.2 [72 to 100] | 91.3 [68 to 100]
  Time-compressed (50%) speech in quiet | 95.7 [60 to 100] | 96.4 [84 to 100] | 86.4 [24 to 100]
  Time-compressed (50%) speech in noise | 89.5 [72 to 100] | 80.2 [60 to 96] | 57.9 [8 to 92]
  Time-compressed (66%) speech in quiet | 92.8 [60 to 100] | 86.4 [52 to 100] | 66.9 [24 to 100]
  Time-compressed (66%) speech in noise | 47.7 [8 to 80] | 26.2 [4 to 60] | 11.3 [0 to 44]
  Time-compressed (80%) speech in quiet | 39.8 [8 to 88] | 12.2 [0 to 60] | 7.1 [0 to 64]
  Time-compressed (80%) speech in noise | 1.4 [0 to 8] | 0.7 [0 to 4] | 0.3 [0 to 4]
  Interrupted (50%) speech in quiet | 98.5 [88 to 100] | 96.2 [80 to 100] | 85.6 [56 to 100]
  Interrupted (50%) speech in noise | 89.7 [68 to 100] | 84.7 [64 to 100] | 58.7 [20 to 92]
  Interrupted (66%) speech in quiet | 98.3 [88 to 100] | 94.9 [80 to 100] | 73.3 [24 to 100]
  Interrupted (66%) speech in noise | 69.8 [40 to 84] | 60.7 [24 to 84] | 36.6 [8 to 84]
  Interrupted (80%) speech in quiet | 86.3 [60 to 100] | 70.7 [8 to 92] | 46.1 [4 to 96]
  Interrupted (80%) speech in noise | 47.1 [20 to 84] | 38.9 [4 to 60] | 19.7 [0 to 64]
  Time-compressed/Expanded (50%) speech in quiet | 98.5 [84 to 100] | 96.7 [88 to 100] | 86.3 [36 to 100]
  Time-compressed/Expanded (50%) speech in noise | 93.4 [84 to 100] | 86.9 [56 to 100] | 69.1 [32 to 100]
  Time-compressed/Expanded (66%) speech in quiet | 98 [72 to 100] | 95.6 [80 to 100] | 77.4 [40 to 100]
  Time-compressed/Expanded (66%) speech in noise | 83.7 [40 to 100] | 72.7 [24 to 92] | 50.7 [10 to 96]
  Time-compressed/Expanded (80%) speech in quiet | 93.7 [64 to 100] | 89.5 [56 to 100] | 66 [24 to 100]
  Time-compressed/Expanded (80%) speech in noise | 75.7 [40 to 100] | 57.6 [32 to 76] | 30 [4 to 76]

ADVERSE EVENTS:
Time Frame: over the course of up to three 2-hour visits, spaced an average of one week apart
Description: Sounds presented at a potentially damaging level
Arm/Group | Younger Normally-hearing Listeners | Older Normally-hearing Listeners | Hearing-impaired Listeners
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes